CLINICAL TRIAL: NCT07308626
Title: Acute Effects of Reformer, Cadillac, and Chair Pilates Appa-ratuses on Cardiac Autonomic Modulation and Flexibility in Sedentary Middle-Aged Women
Brief Title: Acute Effects of Reformer, Cadillac, and Chair Pilates Appa-ratuses on Cardiac Autonomic Modulation and Flexibility
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Princess Nourah Bint Abdulrahman University (Other)
Responsible Party: Principal Investigator, Monira Aldhahi, Associate Prof, Princess Nourah Bint Abdulrahman University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: PNU-8
Record Dates: First submitted 2025-12-09; First posted 2025-12-29 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Healhty

STUDY DESIGN:
Intervention Model Description: This study uses a randomized, counterbalanced crossover design in which all participants complete three separate Pilates exercise sessions performed on different apparatuses (reformer, cadillac, and chair). Each participant experiences all interventions in a rotating order to minimize sequence effects. The crossover model allows each participant to serve as her own control, improving the ability to detect differences in acute physiological responses between apparatus types
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Reformer Pilates Session (Experimental): Participants complete a single 50-minute Pilates session on a reformer apparatus using standardized beginner-level exercises. All movements are performed under instructor supervision. This arm is part of a randomized crossover design in which all participants complete all three apparatus conditions.
  Interventions: Behavioral: Reformer-based Pilates
- Cadillac Pilates Session (Experimental): Participants complete a single 50-minute Pilates session on a cadillac apparatus using standardized beginner-level exercises. This arm is one condition within the randomized crossover design, and all participants perform this and the other apparatus sessions.
  Interventions: Behavioral: Cadillac-based Pilates
- Chair Pilates Session (Experimental): Participants complete a single 50-minute Pilates session on a Pilates chair apparatus using standardized beginner-level exercises. All participants complete this arm as part of the crossover structure.
  Interventions: Behavioral: Chair Pilates Session

INTERVENTIONS:
Behavioral: Reformer-based Pilates — A supervised 50-minute Pilates exercise session performed on the reformer apparatus. Participants complete standardized beginner-level movements using spring resistance. The session emphasizes controlled full-body movement and postural stability.
  Arms: Reformer Pilates Session
Behavioral: Cadillac-based Pilates — A supervised 50-minute Pilates session using the cadillac apparatus. Participants perform beginner-level exercises incorporating bars and spring systems to support controlled movement patterns targeting the upper and lower body.
  Arms: Cadillac Pilates Session
Behavioral: Chair Pilates Session — A supervised 50-minute Pilates session performed on a Pilates chair apparatus. Participants complete a series of standardized beginner-level exercises using spring resistance to train core control, lower-limb strength, and stability.
  Arms: Chair Pilates Session

SUMMARY:
This study looked at how different types of Pilates equipment affect heart function and flexibility right after exercise in sedentary middle-aged women. Pilates can be performed on several apparatuses, such as the reformer, cadillac, and chair, and each device places different demands on the body. However, it is not well known whether these differences lead to different short-term effects on the heart or on flexibility.

In this study, 15 women completed three separate Pilates sessions-one on each apparatus-on different days. During every session, researchers measured heart rate variability (a way to assess how the heart responds to and recovers from exercise). Flexibility was also tested before and after each session.

This information may help instructors and clinicians choose the most appropriate Pilates equipment based on individual goals.

DETAILED DESCRIPTION:
Pilates is widely used to improve strength, posture, and flexibility, and it may also influence how the heart responds to exercise. Many Pilates programs use equipment such as the reformer, cadillac, and chair, which provide adjustable spring resistance and allow movement in different body positions. Although these apparatuses are commonly used in fitness and rehabilitation settings, little is known about whether they create different short-term effects on cardiovascular function or flexibility, especially in people who are sedentary.

This study designed to compare the immediate effects of three Pilates apparatuses-reformer, cadillac, and chair-on heart rate variability (a marker of cardiac autonomic activity) and flexibility in sedentary middle-aged women. Understanding these effects may help practitioners choose equipment that best supports specific goals, such as improving cardiovascular recovery or increasing muscle flexibility.

Each participant will complete one exercise session on each apparatus in a randomized order. Heart rate variability will be measured before exercise, during exercise, and throughout a short recovery period to observe how the body responded and returned to a resting state. Flexibility will be assessed before and after each session to determine the immediate physical benefit of the different apparatus types.

This study may help clarify whether specific Pilates equipment provides unique physiological advantages. Such information may support more targeted exercise prescriptions for individuals who are beginning Pilates, those with limited fitness experience, or those seeking improvements in flexibility or cardiovascular regulation.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Age 40 to 60 years
* Sedentary (not engaged in regular physical activity)
* No prior experience with Pilates apparatus-based exercise
* Able to provide informed consent

Exclusion Criteria:

* Known metabolic or cardiovascular disease
* Regular use of medications that influence heart rate or autonomic function
* Current smoker
* Musculoskeletal injuries or limitations that prevent safe participation in exercise
* Any condition that, in the opinion of the investigators, would interfere with study participation or data collection

Ages: 40 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2025-07-25 (Actual); Primary Completion 2025-09-25 (Actual); Study Completion 2025-10-25 (Actual)

PRIMARY OUTCOMES:
Heart Rate Variability (HRV) | Pre-exercise; during exercise; 10, 20, 30, and 40 minutes post-exercise
  Heart rate fluctuations are measured using a chest-strap heart rate monitor to evaluate cardiac autonomic modulation. The measurements include the average time between heartbeats, the root mean square of differences between successive heartbeats, and the standard deviation of normal heartbeat intervals. These values are analyzed using specialized heart rhythm analysis software. Increases or decreases in these values reflect changes in autonomic nervous system activity. This outcome is used to compare acute cardiovascular responses between the different Pilates apparatus sessions.

SECONDARY OUTCOMES:
Flexibility (Sit-and-Reach Test) | Pre-exercise; immediately post-exercise; 40 minutes post-exercise
  Flexibility is assessed using a standardized sit-and-reach box. Participants perform two trials, and the best score (in centimeters) is recorded. This measure evaluates immediate and short-term changes in lower-back and hamstring flexibility after each apparatus session.

CONTACTS AND LOCATIONS:
Locations (1):
- Bursa Uludag University, Bursa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided